CLINICAL TRIAL: NCT03552822
Title: Clinical Outcomes in Patients Undergoing Cesarean Section Via the Enhanced Recovery After Surgery (ERAS) Pathway: a Retrospective Study
Brief Title: Cesarean Section Via Enhanced Recovery
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mark Powell, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 45678910
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Results first posted 2022-03-07 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS Implemented Group: Enhanced recovery after surgery (ERAS) protocol implementation for patients undergoing cesarean delivery.
  Interventions: Other: ERAS Protocol Implementation
- Pre-ERAS - Non-ERAS Implemented Group: Non-Enhanced recovery after surgery (ERAS) protocol implementation for patients undergoing cesarean delivery.

INTERVENTIONS:
Other: ERAS Protocol Implementation — Implementation of ERAS Protocol Implementation
  Groups: ERAS Implemented Group

SUMMARY:
Enhanced Recovery After Surgery (ERAS) protocols have been proven to be very successful in specific patient populations. An example is with ERAS for colorectal surgery. ERAS protocols in this patient population have been shown to reduce overall morbidity and hospital length of stay (LOS). At the University of Alabama at Birmingham (UAB), the institution has had successful implementation of ERAS protocols for several surgical specialties including colorectal, breast, spine, gynecology, and gynecology-oncology. However, the institution currently does not have a protocol in place for the most commonly performed surgical procedure - cesarean delivery. At UAB, the institution performs approximately 1,000 cesarean deliveries per year.

The investigators believe that an ERAS protocol will be beneficial for these patients. Currently, there is very little data published on ERAS protocols. Although this patient population is ideal for an ERAS protocol, there are several barriers that have to be overcome. The data published show promising results for ERAS protocols with cesarean delivery. A larger tertiary care center showed earlier discharge with lower re-admission rates with an ERAS pathway.

Currently, the investigators have created a multidisciplinary group at UAB to establish an ERAS protocol for patients undergoing cesarean delivery. This group includes anesthesiologists, obstetricians, nursing, neonatology, pharmacy, and informatics. Once the investigators have implemented this protocol, the investigators would like to perform a retrospective analysis to determine if there are any significant changes in our desired outcomes the investigators will study. Our goal is to demonstrate significantly improved outcomes in the investigators' measured endpoints. The investigators believe that this information will be very useful because although there is a national interest in creating ERAS protocols for cesarean deliveries, there currently is very little published on the subject. The investigators would like to publish the investigators' results and protocol as a resource for other institutions to adopt.

DETAILED DESCRIPTION:
The investigators are implementing an enhanced recovery after surgery (ERAS) protocol for patients undergoing cesarean delivery. The purpose of the ERAS protocol is to optimize care provided to patients (patient education, nutrition, pain management, early ambulation, etc.). The anticipated date of protocol initiation is May 2018. Once this protocol has been in place for approximately 6 months to one year, the investigators would like to retrospectively review data on these patients and compare outcomes to a similarly-matched group of patients the year preceding protocol implementation. Specific outcomes the investigators will assess are: hospital length of stay, post-operative pain scores, opioid consumption, patient satisfaction [through IRB-approved survey (protocol X300001121)], surgical site infection rates, readmission rates, and unscheduled clinic and maternal evaluation unit (MEU) visits before the first scheduled postpartum visit. The investigators also plan to track compliance monthly with the adherence to the protocol. Since the investigators want to track compliance (both as a quality improvement project as well as research), the investigators are requesting (Institutional Review Board) IRB approval now.

ELIGIBILITY:
Inclusion Criteria:

Any patient 18 years or older whom is scheduled for an elective cesarean section from one of the participating clinics: Prime Care, Maternal Fetal Medicine (MFM), Obstetrics Complications Clinic (OBCC).

Exclusion Criteria:

1. Age less than 18 years old;
2. urgent or emergent cesarean delivery;
3. diagnosis of preeclampsia;
4. coagulopathy that contraindicates neuraxial block placement;
5. abnormal placentation;
6. opioid abuse disorder;
7. type C diabetic or greater.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on gender identity
Study Population: Patients 18 years or older whom is scheduled for an elective cesarean section from one of the participating clinics: Prime Care, MFM, OBCC.
Sampling Method: Non-Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Lester, MD, Study Chair — UAB Department of Anesthesiology, Critical Care Division
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
Started | 112 | 429
Completed | 112 | 429
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group | Total
Number analyzed (Participants) | 112 | 429 | 541
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.79 (4.96) | 30.58 (5.76) | 30.42 (5.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 429 | 541
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 10 | 13
  Black or African American | 46 | 181 | 227
  Hispanic or Latino | 13 | 54 | 67
  White | 38 | 121 | 159
  Other | 5 | 40 | 45
  Decline/Unknown/Missing | 7 | 23 | 30
Region of Enrollment [Number; unit: participants]
  United States | 112 | 429 | 541
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI was missing for 7 participants (3 in the ERAS Implemented group, 4 in pre-ERAS group)
  kg/m^2
    number analyzed (Participants) | 109 | 425 | 534
    (all) | 36.73 (7.84) | 35.09 (14.26) | 35.43 (13.22)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Measurement of opioid consumption in oral morphine equivalents
Time Frame: From 1 to 72 hours post surgery
Measure: Mean (Standard Error); unit: oral morphine equivalents (mg)
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
Number analyzed (Participants) | 112 | 429
oral morphine equivalents (mg) | 60.34 (4.82) | 104.33 (4.92)
Statistical Analysis 1: Comparison: ERAS Implemented Group vs Pre-ERAS - Non-ERAS Implemented Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Overall Average Pain Scores
Description: Pain scores post-cesarian section will be obtained using clinical data gathered by the care team providing routine clinical care, and asking routine pain score questions. The scale used is the standard 1-10 pain scale, with 1 being no pain or very mild discomfort, and 10 being very severe pain. Thus, higher values indicate a worse outcome. For each subject, pain scores obtained during the 72 hours post-surgery will be averaged to obtain an overall average pain score.
Time Frame: From 1 to 72 hours post surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
Number analyzed (Participants) | 112 | 429
score on a scale | 1.61 (0.13) | 1.90 (0.07)
Statistical Analysis 1: Comparison: ERAS Implemented Group vs Pre-ERAS - Non-ERAS Implemented Group; Test type: Superiority; p = 0.037, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Ambulation
Description: Length of time between surgery and first recorded ambulation. A total of 9 patients are missing data in the electronic medical record and this was accounted for in our analysis but are not represented in the numbers below.
Time Frame: From 1 to 72 hours post surgery
Measure: Mean (Standard Error); unit: hours
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
Number analyzed (Participants) | 108 | 424
hours | 9.76 (0.69) | 32.89 (1.23)
Statistical Analysis 1: Comparison: ERAS Implemented Group vs Pre-ERAS - Non-ERAS Implemented Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Oral Intake
Description: Time to first oral intake of clear liquids. A total of 9 patients are missing data in the electronic medical record and this was accounted for in our analysis but are not represented in the numbers below.
Time Frame: From 1 to 24 hours post surgery
Measure: Mean (Standard Error); unit: hours
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
Number analyzed (Participants) | 108 | 424
hours | 2.19 (0.07) | 3.58 (0.09)
Statistical Analysis 1: Comparison: ERAS Implemented Group vs Pre-ERAS - Non-ERAS Implemented Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Postoperative Nausea and Vomiting
Description: Treatment for postoperative nausea and vomiting was assessed using the total amount of ondansetron given postoperatively.
Time Frame: From 1 to 72 hours post surgery
Measure: Mean (Standard Error); unit: milligrams (mg)
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
Number analyzed (Participants) | 112 | 429
milligrams (mg) | 1.82 (0.28) | 1.48 (0.14)
Statistical Analysis 1: Comparison: ERAS Implemented Group vs Pre-ERAS - Non-ERAS Implemented Group; Test type: Superiority; p = 0.108, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Readmission Rates
Description: Readmissions to the hospital
Time Frame: Up to 21 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
Number analyzed (Participants) | 112 | 429
Participants | 3 | 4
Statistical Analysis 1: Comparison: ERAS Implemented Group vs Pre-ERAS - Non-ERAS Implemented Group; Test type: Superiority; p = 0.159, Fisher Exact

7. Secondary Outcome: Foley Catheter Removal
Description: Time to Foley catheter removal postoperative. A total of 9 patients are missing data in the electronic medical record and this was accounted for in our analysis but are not represented in the numbers below.
Time Frame: From 1 to 24 hours post surgery
Measure: Mean (Standard Error); unit: hours
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
Number analyzed (Participants) | 108 | 424
hours | 11.29 (0.71) | 21.17 (0.40)
Statistical Analysis 1: Comparison: ERAS Implemented Group vs Pre-ERAS - Non-ERAS Implemented Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Postoperative Temperature
Description: Temperature recorded in post-anesthesia care unit. A total of 9 patients are missing data in the electronic medical record and this was accounted for in our analysis but are not represented in the numbers below.
Time Frame: 1 hour post surgery
Measure: Mean (Standard Error); unit: degrees Fahrenheit
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
Number analyzed (Participants) | 108 | 424
degrees Fahrenheit | 97.54 (0.07) | 97.37 (0.02)
Statistical Analysis 1: Comparison: ERAS Implemented Group vs Pre-ERAS - Non-ERAS Implemented Group; Test type: Superiority; p = 0.020, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Hospital Length of Stay
Description: Length of stay in hospital post-cesarian. A total of 9 patients are missing data in the electronic medical record and this was accounted for in our analysis but are not represented in the numbers below.
Time Frame: Time of admission until time of discharge, generally not over one week
Measure: Mean (Standard Error); unit: hours
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
Number analyzed (Participants) | 108 | 424
hours | 81.37 (1.85) | 90.76 (2.25)
Statistical Analysis 1: Comparison: ERAS Implemented Group vs Pre-ERAS - Non-ERAS Implemented Group; Test type: Superiority; p = 0.085, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 30 days postoperative
Arm/Group | ERAS Implemented Group | Pre-ERAS - Non-ERAS Implemented Group
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/429
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/429
Other Adverse Events (participants affected / at risk) | 0/112 | 0/429

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03552822/Prot_SAP_001.pdf